CLINICAL TRIAL: NCT03833284
Title: Implementation of a Transvaginal Ultrasound Surveillance Program in Women With a History of Previous Preterm Birth: Disseminating Evidenced Based Practices for Reducing Preterm Birth in Appalachian Kentucky
Brief Title: Transvaginal Ultrasound: Preterm Birth Prevention in Appalachia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Niraj Chavan (Other)
Responsible Party: Sponsor-Investigator, Niraj Chavan, Assistant Professor in Maternal Fetal Medicine, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 45131
Record Dates: First submitted 2019-01-03; First posted 2019-02-06 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Preterm Birth
Keywords: Transvaginal Ultrasound; Telemedicine
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participant Barriers to TVU Screening (Experimental): Patients with a history of pre-term birth will be identified through a review of their medical history. Patients will then be asked to complete a survey assessing their knowledge of transvaginal ultrasound screening. Patients will then be asked to attend in-person or online workshops designed to increase patient knowledge of TVU screening guidelines and benefits. Finally, patients will complete exit surveys to determine whether their attitudes and beliefs towards screening have changed over time.
  Interventions: Behavioral: Participant Barriers to TVU Screening
- Provider Barriers to TVU Screening (Experimental): Obstetric and Gynecologic Providers will be identified based on prior working relationships with the University of Kentucky outreach programs. Chosen providers will be asked to complete a survey assessing their attitudes towards TVU screening. Following completion, providers will be asked to attend either in-person or online workshops designed to increase provider knowledge of TVU screening guidelines and benefits. Finally, providers will complete exit surveys to determine whether their attitudes and beliefs toward screening have changed over time.
  Interventions: Behavioral: Provider Barriers to TVU Screening

INTERVENTIONS:
Behavioral: Participant Barriers to TVU Screening — Workshops tailored toward patients to increase knowledge about TVU screening guidelines and benefits.
  Arms: Participant Barriers to TVU Screening
Behavioral: Provider Barriers to TVU Screening — Workshops tailored toward providers to increase knowledge about TVU screening guidelines and benefits.
  Arms: Provider Barriers to TVU Screening

SUMMARY:
Preterm Birth is the number one cause of infant morbidity and mortality worldwide and represents an important health disparity in the United States, particularly across the state of Kentucky. The best biomarker for the prediction of preterm birth is transvaginal ultrasound (TVU). This study will attempt to identify and rectify provider and patient related barriers to TVU screening implementation.

DETAILED DESCRIPTION:
Preterm birth is the number one cause of infant morbidity and mortality worldwide and represents an important health disparity in the United States, and especially across the state of Kentucky. The best biomarker for the prediction of preterm birth is transvaginal ultrasound (TVU) measurement of cervical length. However, several unique provider and patient related barriers for implementation of this screening limit the widespread uptake of this evidence based practice in Appalachian KY. The investigators propose to adopt a dissemination and implementation science approach using the Consolidated Framework for Implementation Research (CFIR) as the guiding framework for identification of key areas of knowledge deficits as well as attitudes, practices and perceived barriers among prenatal care providers and patients in eastern KY towards TVU cervical length screening using a mixed - methods design. This will be utilized to develop a multifaceted implementation strategy best suited for addressing and overcoming barriers identified by the target population in eastern KY. The investigators anticipate that such an implementation strategy will likely include an educational component targeting obstetric care providers and patients in addition to hands-on TVU cervical length evaluation as well as telemedicine support and surveillance. Three community based sites (Hazard, Morehead and Ashland, KY) will be recruited for implementation of this multi-component pilot program focused on community engagement and outreach targeting obstetric providers and their patients. At the end of the pilot implementation phase, acceptability of the study intervention and feasibility of implementation will be evaluated along with a preliminary assessment of effectiveness of implementation.

ELIGIBILITY:
Inclusion Criteria: Participant

* Female Sex
* Prior history of preterm birth (for initial set of interviews), no preterm birth history required for intervention feedback
* Current pregnant status

Exclusion Criteria: Participant

* Male Sex

Inclusion Criteria: Provider

* Certified as obstetric/gynecologic provider

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Change in attitudes towards TVU screening among patients and practitioners | At baseline and at one year.
  The primary purpose of this study is to evaluate the change in attitudes towards TVU screening among patients and practitioners. This will be accomplished by conducting a qualitative interview with each participant at baseline and again at one year (after completing the CLEAR program workshop).
Potential for future TVU screening implementation based on changes in attitudes towards TVU screening among providers and participants. | At baseline and at one year.
  The primary purpose of this study is to evaluate the change in attitudes towards TVU screening among patients and practitioners. This will be accomplished by conducting a qualitative interview with each participant at baseline and again at one year (after completing the CLEAR program workshop). Analysis of these interviews will aid in determining feasibility of implementing a future TVU screening component in Obstetric and Gynecologic care.

SECONDARY OUTCOMES:
Rate of preterm birth at <34 weeks gestation | Through study completion, average of 1 year from study initiation
  Subjects (patients) included in this study will be followed to determine rate of preterm birth at various time points.
Rate of preterm birth at <37 weeks gestation | Through study completion, average of 1 year from study initiation
  Subjects (patients) included in this study will be followed to determine rate of preterm birth at various time points.
Number of TVU scans identifying a short cervix (≤ 25 mm) in any pregnant women at each study site | Through study completion, average of 1 year from study initiation.
  Records of TVU scans identifying a short cervix among the study population will be analyzed to determine the rate of short cervix issues among the population. The percentage will aid in determining the need for future TVU screening in similar populations.
Rate of inpatient hospitalization for preterm labor management prior to delivery | Through study completion, average of 1 year from study initiation.
  Subjects (patients) included in this study will be followed to determine whether they are subjects to hospitalization prior to birthing due to complications associated with preterm labor.
Rates of clinical therapy | Through study completion, average of 1 year from study initiation.
  Defined as prescribing vaginal progesterone or performing cervical cerclage

CONTACTS AND LOCATIONS:
Overall Officials: Niraj Chavan, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No